CLINICAL TRIAL: NCT02163486
Title: The Influence of Head and Neck Position On The Oropharyngeal Leak Pressure of LMA Unique ™ and I-GEL™
Brief Title: Comparison Between the I-gel and the LMA-Unique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Sule Ozbilgin, Anaesthesiology and Reanimation, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 10-11.1/30
Record Dates: First submitted 2014-06-10; First posted 2014-06-13 (Estimated); Results first posted 2018-10-19 (Actual); Last update posted 2018-10-19 (Actual); Status verified 2017-12

CONDITIONS: Anaesthesia
Keywords: I-gel; oropharyngeal leak pressure; head position

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group U (UNIQUE) (Active Comparator): Group LMA- UNIQUE, inserted according to described standard method. Between 30-40 kg, no.3. Between 50-70 kg, no. 4 Between 70-100 kg, no. 5. LMA-Unique Before SGAD is inserted, a water-based lubricant without local anesthetic, was spread on the surfaces that will touch the palate and LMA-U cuff was completely deflated.oup U (UNIQUE): Group Laryngeal Mask Airway-Unique.
  Interventions: Device: Group U (UNIQUE)
- Group I (I-GEL ): Group I-GEL (Experimental): Group I (I-GEL): Between 30-60 kg, no. 3. Between 50-90 kg, no. 4. For > 90 kg no.5. I-GEL
  Interventions: Device: I-GEL

INTERVENTIONS:
Device: Group U (UNIQUE) — Before LMA-Unique was inserted, to lubricate the surface in contact with the palate a water-based gel without local anesthetic was applied to completely cover the LMA-Unique cuff.
  Other Names: Laryngeal Mask Airway-Unique; Teleflex, The Laryngeal Mask Company Limited, Singapore .
  Arms: Group U (UNIQUE)
Device: I-GEL — Before I-gel was inserted, to lubricate the surface in contact with the palate a water-based gel without local anesthetic was applied to completely cover the I-GEL cuff.
  I-GEL: K-Y Jelly® is a registered trademark of Johnson and Johnson Inc
  Other Names: Group I (I-GEL): I-GEL
  Arms: Group I (I-GEL ): Group I-GEL

SUMMARY:
Airway management is one of the basic topics in anesthetic practice. Use of endotracheal intubation and face mask are standard methods to maintain an open airway widely adopted for many years. As a result of a search for more appropriate choices from the point of view of effectiveness, reliability and side effects, supraglottic airway devices (SGAD) have been developed.

SGAD's are used for thyroid surgery, ear surgery, carotid endarterectomy, adenotonsillectomy and laser pharyngoplasty, which require a variety of head-neck positions. Changing the head and neck position leads to changes in the shape of the pharynx, which causes variation in the cuff pressure and oropharyngeal leak pressure. Oropharyngeal leak pressure values play a determining role in protecting the airway from high cuff pressure. Additionally it shows that the laryngeal mask is correctly placed and is a sign of the effectiveness of positive pressure ventilation. During surgery head-neck and trunk position may change. As a result there is a need for research evaluating the effect of head and neck position on oropharyngeal leak pressure during SGAD use.

AIM

The aim of this study is to compare the effect of different head and neck positions on the oropharyngeal leak pressure in LMA-Unique and I-Gel applications. Additionally the placement duration, ease and success of these two supraglottic airway devices will be compared.

DETAILED DESCRIPTION:
This prospective, randomized, double-blind study will receive permission from the Local Research Ethics Committee and after obtaining patients' informed consent, 103 patients with American society of anesthesiologists (ASA) classification group I-II, between 18-65 years, undergoing elective surgery with indications for supraglottic airway device placement were included in the study.

All patients preoperatively evaluated and ASA and Mallampati classification recorded.

All SGAD's inserted by the same experienced researcher. After placement of laryngeal mask, to standardize postoperative pharyngeal morbidity, cuff pressure (cuff pressure manometer, Ruch, Germany) was monitored.

EXCLUSION CRITERIA:

* Any neck or upper respiratory pathology
* Those at risk of gastric content regurgitation/aspiration (previous upper Gastro-intestinal surgery, known hiatus hernia, Gastroesophageal reflux, history of peptic ulcer, full stomach, pregnancy)
* Possibility of and those with history of difficult intubation (history of impossible intubation, Mallampati classification 3-4, sterno mental distance less than 12 cm, thyromental distance less than 6 cm, head extension less than 90 degrees, mouth opening less than 1.5 cm)
* Those with low pulmonary compliance or high airway resistance (morbid obesity, lung disease)
* Throat pain, dysphagia and dysphonia
* Patients with cervical disc hernia

Patients taken to the operating room were given standard monitoring before anesthesia induction. Patients were preoxygenated with 6 L/min oxygen for 3 minutes through a face mask.

Anesthesia induction was provided by 0.02 mg/kg midazolam, 1-2 mcg/kg fentanyl, 1.5-2 mg/kg propofol and 0.5 mg/kg rocuronium.

All patients have neuromuscular junction monitoring (TOF-GUARD, Biometer International A.S. DENMARK) and when TOF is zero SGAD was inserted with the standard method according to the firm's recommendations.

During SGAD placement, if necessary additional dose of 0.5 mg/kg propofol was given depending on patient reaction. During this procedure cases were ventilated with 100% oxygen though a mask.

STUDY GROUPS:

Group U (UNIQUE): LMA- UNIQUE, inserted according to described standard method

Group I (I-GEL ) : I-GEL, inserted with standard technique according to users manual

For LMA-U the laryngeal mask cuff was inflated so that cuff pressure is less than 60 cm H2O with leak preventive volume. After the operation before the laryngeal mask was removed the cuff pressure was measured again and recorded.

To check SGAD placement bilateral chest movement was observed and capnography be used to confirm a square wave shape. After SGAD was placed oropharyngeal leak test was completed. Oropharyngeal leak pressure were tested in both groups first in neutral head position, then at maximum extension and with head at maximum rotation to the right. In every position the leak measurement was made 60 seconds after position is changed. In order to prevent the SGAD from being seen by the researcher during the tests the patient's head was covered.

Oropharyngeal leak pressure was measured with the ring system expiratory valve closed and 4 L/min flow. To prevent exposure of the lungs to barotrauma, when peak airway pressure reaches 40 cm H2O the expiratory valve was opened .

Leak pressure was evaluated in two ways;

1. The stethoscope is placed above the patient's left thyroid part of the trachea and the sound of a leak is listened for
2. Checked when the aneroid manometer is held steady (manometer stability test)

When the sound of the leak is heard, the pressure on the manometer were recorded separately in both situations.

Anesthesia was maintained with 5% O2/air mix with 1.5-2.5% sevoflurane. Systolic arterial pressure (SAP), diastolic arterial pressure (DAP), mean arterial pressure (MAP), and heart rate (HR) values were measured and recorded immediately before anesthesia induction, immediately before airway device placement and at 1, 2, and 3 minutes after airway placement is checked. The time for successful placement (duration from mouth opening to first successful ventilation), number of attempts, and ease of placement were recorded.

Ease of insertion:

1. no reaction
2. straining, retching
3. alternative airway management

The Mallampati score, type of supraglottic airway device, type of operation and total duration of anesthesia were recorded. Any problems occurring during head and neck positions was noted.

The cuff pressure was measured after surgery while the patient is still in deep anesthesia.

When the patient is conscious the SGAD was removed and the duration of use was recorded (time from insertion to removal).

After the SGAD is removed the presence of blood was evaluated

1. no blood
2. trace amounts of blood
3. definite amount of blood

The patients throat pain, voice loss and difficulty swallowing were evaluated when leaving the recovery room and by telephone 24 hours later by a researcher blind to the insertion technique. To evaluate throat pain the VAS 10 (verbal analogue scale) was used

EXPULSION CRITERIA:

* Oxygen saturation by pulse oximetry values falling by 90% during airway insertion
* Cases developing laryngospasm
* Cases with incomplete records

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II
* 18-65 years

Exclusion Criteria:

* Any neck or upper respiratory pathology
* Those at risk of gastric content regurgitation/aspiration (previous upper gastro-intestina system surgery, known hiatus hernia, gastroesophageal reflux, history of peptic ulcer, full stomach, pregnancy)
* Possibility of and those with history of difficult intubation (history of impossible intubation, Mallampati classification 3-4, sterno mental distance less than 12 cm, thyromental distance less than 6 cm, head extension less than 90 degrees, mouth opening less than 1.5 cm)
* Those with low pulmonary compliance or high airway resistance (morbid obesity, lung disease)
* Throat pain, dysphagia and dysphonia
* Patients with cervical disc hernia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2010-12; Primary Completion 2011-02 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: FARUK ÖZATA, M.D., Principal Investigator — STUDY DESİGN; BAHAR KUVAKİ, M.D., Study Director — Dokuz Eylül University, School of Medicine, Department of Anesthesiology and Reanimation
Locations (1):
- Dokuz Eylül University, School of Medicine, Department of Anesthesiology and Reanimation, Izmir, Narlıdere, Turkey (Türkiye)

RESULTS

PARTICIPANT FLOW:
Groups:
- Group U (UNIQUE): Group LMA- UNIQUE, inserted according to described standard method. Between 30-40 kg, no.3. Between 50-70 kg, no. 4 Between 70-100 kg, no. 5. LMA-Unique Before LMA-U is inserted, a water-based lubricant without local anesthetic, was spread on the surfaces that will touch the palate and LMA-Unique cuff was completely deflated. Group U (UNIQUE): Group Laryngeal Mask Airway-Unique.
  Group U (UNIQUE): Before LMA-Unique was inserted, to lubricate the surface in contact with the palate a water-based gel without local anesthetic was applied to completely cover the LMA-Unique cuff.
- Group I (I-GEL ): Group I-GEL: Group I (I-GEL): Between 30-60 kg, no. 3. Between 50-90 kg, no. 4. For > 90 kg no.5. I-GEL
  I-GEL: Before I-gel was inserted, to lubricate the surface in contact with the palate a water-based gel without local anesthetic was applied to completely cover the I-GEL cuff.
  I-GEL: K-Y Jelly® is a registered trademark of Johnson and Johnson Inc
Period: Overall Study
Arm/Group | Group U (UNIQUE) | Group I (I-GEL ): Group I-GEL
Started | 51 | 52
Completed | 50 | 50
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group U (UNIQUE) | Group I (I-GEL ): Group I-GEL | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 50 | 50 | 100
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 25 | 48
  Male | 27 | 25 | 52
Region of Enrollment [Number; unit: participants]
  Turkey | 50 | 50 | 100

OUTCOME MEASURES:

1. Primary Outcome: Oropharyngeal Leak Pressure
Description: The aim of this study is to compare the effect of different head and neck positions on the oropharyngeal leak pressure in LMA-Unique and I-Gel applications. Head and neck positions are limited to neutral, extension and right laterally deviated.
Time Frame: Immediately after head and neck positioning is completed
Measure: Mean (Standard Deviation); unit: cm H20
Arm/Group | Group U (UNIQUE) | Group I (I-GEL ): Group I-GEL
Number analyzed (Participants) | 50 | 50
cm H20
  when neutral position | 25.06 (7.53) | 28.24 (8.29)
  when extension position | 22.88 (7.83) | 26.62 (8.77)
  when right position | 27.30 (7.23) | 26.04 (8.61)

2. Secondary Outcome: The Time for Successful Placement (Second)
Description: Duration from mouth opening to first successful ventilation, in seconds
Time Frame: Baseline to first successful ventilation, in seconds
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Group U (UNIQUE) | Group I (I-GEL ): Group I-GEL
Number analyzed (Participants) | 50 | 50
seconds | 13.46 (2.60) | 12.14 (4.22)

3. Secondary Outcome: Number of Attempts
Description: The number of attempts until succesful placement of airway device
Time Frame: Baseline to first successful ventilation,
Population: The number of patients with succesful placement of airway device at the first attempt
Measure: Count of Participants; unit: Participants
Arm/Group | Group U (UNIQUE) | Group I (I-GEL ): Group I-GEL
Number analyzed (Participants) | 50 | 50
Participants
  Succesful First Attempt | 48 | 48
  Succesful second Attempt | 2 | 1
  Succesful third Attempt | 0 | 1

4. Secondary Outcome: Ease of Placement
Description: Ease of placement:
  1. no reaction
  2. straining, retching
Time Frame: Baseline
Measure: Number; unit: participants
Arm/Group | Group U (UNIQUE) | Group I (I-GEL ): Group I-GEL
Number analyzed (Participants) | 50 | 50
participants
  no reaction | 49 | 49
  straining, retching | 1 | 1

5. Secondary Outcome: Incidence of Post-operative Sore Throat
Description: Patients were asked about the presence of sore throat - defined as the presence of constant pain in the throat, voice loss and difficulty swallowing , at postoperative 1st and 24th hours.
Time Frame: at postoperative 1st and 24th hours
Measure: Number; unit: participants
Arm/Group | Group U (UNIQUE) | Group I (I-GEL ): Group I-GEL
Number analyzed (Participants) | 50 | 50
participants | 5 | 0

ADVERSE EVENTS:
Arm/Group | Group U (UNIQUE) | Group I (I-GEL ): Group I-GEL
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No